CLINICAL TRIAL: NCT03004976
Title: Phase 2 Study of Allogeneic Umbilical Cord Blood Infusion for Adults With Ischemic Stroke - CoBIS 2
Brief Title: Study of Allogeneic Umbilical Cord Blood Infusion for Adults With Ischemic Stroke
Acronym: CoBIS 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joanne Kurtzberg, MD (Other)
Collaborators: The Marcus Foundation (Other); Emory University (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Joanne Kurtzberg, MD, Director, Robertson Clinical and Translational Cell Therapy Program, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00077580
Record Dates: First submitted 2016-11-30; First posted 2016-12-29 (Estimated); Results first posted 2022-09-23 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Stroke; Stroke, Acute; Brain Injury, Acute
Keywords: hematopoietic stem cells; umbilical cord blood; stroke; ischemic stroke
MeSH Terms: conditions — Stroke; Brain Injuries; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Umbilical Cord Blood (Experimental): A single intravenous infusion of umbilical cord blood within 3-10 days following stroke.
  Interventions: Biological: Umbilical Cord Blood
- Placebo (Placebo Comparator): A single intravenous infusion of diluent with the same appearance and odor as a cord blood unit within 3-10 days following stroke.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Umbilical Cord Blood — Umbilical cord blood will be infused intravenously through a peripheral IV line after premedication with diphenhydramine, hydrocortisone, and acetaminophen. Units will be from a public cord blood bank with selection based on blood type, race, and the number of cells in the pre cryopreservation product, targeting a dose range of 0.5 to 5 x 10^7 TNCC/kg.
  Other Names: cord blood; hematopoietic stem cells
  Arms: Umbilical Cord Blood
Other: Placebo — The placebo product will be acellular and will consist of tissue culture medium 199 (TC-199 [pink]) with 1% dimethyl sulfoxide (DMSO), which are standard components in cellular products. The volume of placebo product will be 50 mL, which is in the range of a typical UCB unit that has been washed and thawed after cryopreservation. Infusion and premedication procedures will be the same as those conducted for the umbilical cord blood arm.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine the efficacy of a single intravenous infusion of unrelated donor umbilical cord blood (UCB) for improving functional outcomes in patients with ischemic stroke. Eligible subjects will receive an intravenous infusion of UCB or placebo 3-10 days following stroke. Subjects will not receive immunosuppressive or myeloablative medications prior to the infusion. Subjects will be followed for one year post infusion for safety and efficacy. Assessments will examine safety and tolerability of the infusion, change in neurological symptoms, change in quality of life, and emotional and cognitive status. Assessments will occur at 24 hours post infusion, and at 30, 90, 180 and 365 days post infusion.

DETAILED DESCRIPTION:
This is a multicenter, placebo controlled, randomized, double blinded Phase 2 study in 100 subjects 18-90 years of age who have sustained a recent ischemic stroke. Potential subjects can be screened and consented the day of their stroke (Day 1). Treatment with umbilical cord blood (UCB) cells or placebo will be administered intravenously as a single infusion as early as 3 days but no later than 10 days after the patient's stroke. UCB units will be selected from an accredited U.S. public cord bank based on blood type, race and a targeted cell dose ranging between 0.5 to 5 x 10^7 total nucleated cell count (TNCC)/kg. Study subjects will not receive immunosuppressive or myeloablative medications prior to infusion of the cord blood or placebo.

All subjects, families and medical staff will be blinded to treatment arm. When a subject is randomized to study drug at a clinical site without a cord blood bank, the selected cord blood units (CBU) will be shipped frozen overnight to the site. Once selected and available on site, each CBU will be thawed, washed, tested, released and infused intravenously using common standard operating procedures (SOPs) at all sites. For subjects randomized to placebo, a diluent with the same appearance and odor as a CBU will be prepared.

Patients will have baseline magnetic resonance imaging (MRI) and will be assessed at 1, 3, 6, and 12 months for functional outcomes. All patients will receive standard of care therapy while enrolled in this study and all subjects will be strongly encouraged to participate in rehabilitative therapy.

The primary objective of the study is to determine, in a randomized, placebo controlled trial, the efficacy of a single intravenous (IV) infusion of unrelated donor UCB for improving functional outcomes in patients with ischemic stroke. The secondary objectives are as follows:

1. To describe the safety and tolerability of a single IV infusion of unrelated donor UCB in patients with ischemic stroke
2. To evaluate the efficacy of a single IV infusion of unrelated donor UCB for improvement of neurological symptoms following ischemic stroke
3. To evaluate the efficacy of a single IV infusion of unrelated donor UCB for improvement in quality of life and emotional and cognitive status in patients with ischemic stroke

ELIGIBILITY:
Inclusion Criteria:

1. 18-90 years old
2. Recent, acute, cortical, hemispheric, ischemic stroke in the MCA (middle cerebral artery) distribution without a clinically significant midline shift as detected by MRI as a DWI (diffusion-weighted imaging) abnormality. If unable to obtain a MRI scan, patients may be included if there is clear evidence of ischemic cortical involvement in the MCA distribution demonstrated by computed tomography and a clinical exam consistent with cortical involvement.
3. NIHSS 6-15 (R) and 6-20 (L) at the time of informed consent. Subjects with a >4-point increase of NIHSS from time of consent (worsening of score) will not be eligible for infusion.
4. Subjects must have a platelet count >100,000/uL, hemoglobin >8gm/dL, absolute lymphocyte count (ALC) ≥ 1200 for African American patients and ≥1500 for all other racial-ethnic groups, and WBC (white blood cell) count >2,500/uL OR Historical pre-stroke value of ALC ≥ 1200 for African American and ≥1500 for all other racial-ethnic groups within 6 months of stroke

   -And- a post stroke ALC value of ≥ 1000, platelet count >100,000/uL, hemoglobin >8gm/dL and WBC >2,500/uL.
5. Subjects who received tPA (Tissue plasminogen Activator) or underwent endovascular reperfusion may be included in the study
6. Able to provide consent to study or consent is obtained from the patient's legal representative
7. Subjects of childbearing potential must practice effective contraception during the study, and be willing to continue contraception for at least 6 months after intervention so that, in the opinion of the Investigator, they will not become pregnant during the course of the study
8. Is a good candidate for the trial, in the opinion of the Investigator
9. Agrees to participate in follow-up visits
10. ABO/Rh and race matched CBU(s) with a minimum of 0.5 x 10^7 TNCC/kg based on the pre-cryopreservation TNCC is available for infusion
11. Has not had a disease or therapy that would compromise current immune function.
12. Has a serum creatinine ≤2 mg/dL OR Glomerular Filtration Rate (GFR) ≥30mL/min

Exclusion Criteria:

An individual is ineligible to participate if any of the following apply:

Exclusionary Medical Conditions:

1. Medical history of neurological or orthopedic pathology with a deficit as a consequence that results in a modified Rankin Scale >1 before stroke or has a pre existing cognitive deficit
2. Clinically significant and/or symptomatic hemorrhage associated with stroke
3. Evidence of significant midline shift as assessed by CT or MRI who are felt to be at high risk for neurological decompensation or need for decompressive hemicraniectomy due to hemispheric edema
4. New intracranial hemorrhage, edema, or mass effect that may place patient at increased risk for secondary deterioration when assessed prior to infusion
5. Hypotension as defined as the need for IV pressor support of SBP (systolic blood pressure) <90
6. Isolated brain stem stroke
7. Pure lacunar stroke
8. At time of consent, patients who are mechanically ventilated or, at the investigator's discretion are felt to be likely to need mechanical ventilation are excluded.
9. Requires a craniotomy
10. Serious psychiatric or neurological disease which could alter evaluation on functional or cognitive scales
11. Active systemic infection that is felt, at the discretion of the Investigator, to place the patient at increased risk for participation in this study
12. Documentation of human immunodeficiency virus positive (HIV+) status in the medical record
13. Active malignancy within 3 years prior to the start of screening excluding skin cancers other than melanoma
14. Known hypercoagulable state or coagulopathy deficiencies such as Factor V Leiden, Antiphospholipid Syndrome (APC), Protein C, Protein S, anticardiolipin antibody, phospholipid syndrome or Sickle Cell Disease
15. History of or currently active autoimmune disease, or current immunomodulatory therapy or a recipient of immunomodulatory therapy in the past year.
16. Concurrent illness or condition that in the opinion of the Investigator might interfere with treatment or evaluation of safety
17. Current or recent history of alcohol or drug abuse, or stroke associated with drug abuse that Investigator feels may impair therapy or assessments
18. Pregnant as documented by blood test

Prohibited Concomitant or Prior Therapies

1. Patients currently receiving immunosuppressant drugs, not including glucocorticoid taper, topical/inhaled glucocorticoids
2. History of prior transfusion reaction
3. Currently on dialysis
4. Recipient of bone marrow or organ transplant
5. Hepatic insufficiency (bilirubin >2.5mg/dL or transaminases >5x the ULN) Patients with Gilberts syndrome are eligible for study enrollment if other liver function tests are normal, regardless of bilirubin level
6. Previous or current treatment with angiogenic growth factors, cytokines, gene or stem cell therapy
7. Participating in another interventional clinical trial of an investigational therapy within 30 days of consent.

Other Exclusion Criteria

1. Pregnant or lactating women
2. Unable or unwilling to be evaluated for follow-up visits

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2021-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Kurtzberg, MD, Principal Investigator — Duke University
Locations (6):
- United States (6):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Florida Health Shands Hospital, Gainesville, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Houston Methodist, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Umbilical Cord Blood: A single intravenous infusion of umbilical cord blood within 3-10 days following stroke.
  Umbilical Cord Blood: Umbilical cord blood will be infused intravenously through a peripheral IV line after premedication with diphenhydramine, hydrocortisone, and acetaminophen. Units will be from a public cord blood bank with selection based on blood type, race, and the number of cells in the pre cryopreservation product, targeting a dose range of 0.5 to 5 x 10^7 total nucleated cell count (TNCC)/kg.
- Placebo: A single intravenous infusion of diluent with the same appearance and odor as a cord blood unit within 3-10 days following stroke.
  Placebo: The placebo product will be acellular and will consist of tissue culture medium 199 (TC-199 [pink]) with 1% dimethyl sulfoxide (DMSO), which are standard components in cellular products. The volume of placebo product will be 50 mL, which is in the range of a typical UCB (umbilical cord blood) unit that has been washed and thawed after cryopreservation. Infusion and premedication procedures will be the same as those conducted for the umbilical cord blood arm.
Period: Overall Study
Arm/Group | Umbilical Cord Blood | Placebo
Started | 52 | 27
Completed | 39 | 21
Not Completed | 13 | 6
Not completed — Lost to Follow-up | 7 | 5
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Umbilical Cord Blood | Placebo | Total
Number analyzed (Participants) | 52 | 27 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (13.0) | 64.0 (11.1) | 62.2 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 10 | 31
  Male | 31 | 17 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 8
  Not Hispanic or Latino | 46 | 25 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 6 | 19
  White | 35 | 19 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52 | 27 | 79

OUTCOME MEASURES:

1. Primary Outcome: Shift in Modified Rankin Scale (mRS)
Description: The Modified Rankin Score (mRS) is a disability scale with possible scores ranging from 0 to 6, where 6 = death. Since a shift downward in the mRS scale is considered a clinical improvement, shift scores are calculated from baseline to ensure that, for hypothesis testing purposes, larger shift values represent more clinically desirable outcomes.
Time Frame: baseline to 3 months post infusion
Population: Modified Intention To Treat population (participants who have a baseline and 90 day mRS score)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 47 | 26
score on a scale | 1 [0 to 2] | 1 [0 to 2]
Statistical Analysis 1: Comparison: Umbilical Cord Blood vs Placebo; Primary efficacy analysis (mRS shift from baseline to 90 days); Test type: Other; p = 0.71, Wilcoxon (Mann-Whitney) — Wilcoxon Two Sample Test; Wilcoxon Mann-Whitney Odds = 0.9, 95% CI 2-sided [0.53 to 1.55], Standard Error of Mean 0.248
Statistical Analysis 2: Comparison: Umbilical Cord Blood vs Placebo; Additional analysis of the primary endpoint (mRS score at 90 days), adjusted for baseline mRS, baseline NIHSS, and institution; Test type: Other; p = 0.87, Cumulative Logit Proportional Odds Model; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.4 to 2.3], Standard Error of Mean 0.223

2. Secondary Outcome: Number of Infusion Reactions
Time Frame: up to 1 year post infusion
Population: Safety population
Measure: Number; unit: reactions
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 50 | 27
reactions | 13 | 4

3. Secondary Outcome: Number of Product-related Infections
Time Frame: up to 1 year post infusion
Population: Safety population
Measure: Number; unit: infections
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 50 | 27
infections | 0 | 0

4. Secondary Outcome: Number of Alloimmunization Events
Time Frame: up to 1 year post infusion
Measure: Number; unit: events
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 50 | 27
events | 0 | 0

5. Secondary Outcome: Number of Graft vs. Host Disease Events
Time Frame: up to 1 year post infusion
Population: Safety population
Measure: Number; unit: events
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 50 | 27
events | 0 | 0

6. Secondary Outcome: Number of Study Related and Unexpected Adverse Events (AEs)
Time Frame: up to 1 year post infusion
Population: Safety population
Measure: Number; unit: events
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 50 | 27
events | 0 | 0

7. Secondary Outcome: Mortality
Time Frame: up to 1 year post infusion
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 50 | 27
Participants | 4 | 1

8. Secondary Outcome: Number of Participants With Functional Independence
Description: Functional independence at 90 days defined as a 90-day mRS (modified Rankin Scale) score of 0, 1, or 2. The mRS has a range of 0 to 5, where lower scores indicate a better outcome.
Time Frame: 90 days post infusion
Population: Modified Intention To Treat population.
Measure: Count of Participants; unit: Participants
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 47 | 26
Participants | 15 | 6

9. Secondary Outcome: Shift in Modified Rankin Scale (mRS) From Baseline to 30 Days Post Infusion
Description: as for outcome 1
Time Frame: baseline to 30 days post infusion
Population: Modified Intention To Treat population with a 30 day mRS score available
Measure: Median (Inter-Quartile Range); unit: shift in score
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 46 | 25
shift in score | 1 [0 to 1] | 1 [0 to 1]

10. Secondary Outcome: Shift in Modified Rankin Scale (mRS) From Baseline to 180 Days Post Infusion
Description: as for outcome 1
Time Frame: baseline to 180 days post infusion
Population: Modified Intention To Treat population with a 180 day mRS score available
Measure: Median (Inter-Quartile Range); unit: shift in score
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 42 | 24
shift in score | 1 [1 to 2] | 1 [1 to 2]

11. Secondary Outcome: The National Institutes of Health Stroke Scale (NIHSS) Score at 90 Days
Description: The NIHSS has a range of 0 to 42, where higher scores indicate greater impairment.
Time Frame: 90 days post infusion
Population: Modified Intention To Treat population with NIHSS score available
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 41 | 24
score on a scale | 6 [3 to 9] | 6 [3 to 10]

12. Secondary Outcome: Barthel Index (BI) Score at 90 Days
Description: The Barthel Index assesses functional independence, generally in stroke patients. The BI has a range of 0 to 100 with 0 indicating total dependency and 100 indicating complete independence.
Time Frame: 90 days post infusion
Population: Modified Intention To Treat population with BI available at 90 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 43 | 24
score on a scale | 80 [50 to 100] | 85 [45 to 97.5]

13. Secondary Outcome: Stroke Impact Scale-16 (SIS-16) Score at 90 Days
Description: The SIS-16 has a range of 0 to 100 with higher scores indicating a higher quality of life.
Time Frame: 90 days post infusion
Population: Modified Intention to Treat population with SIS-16 score available at 90 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 43 | 24
score on a scale | 59 [42 to 76] | 64 [41.5 to 76.5]

14. Secondary Outcome: The European Quality of Life (EQ-5D-3L) Visual Analogue Score (VAS) at 90 Days
Description: The EQ-5D-3L VAS ranges from 0 to 100 with 0 being the worst possible health status and 100 being the best possible health status.
Time Frame: 90 days post infusion
Population: Modified Intention To Treat population with EQ-5D-3L VAS score available at 90 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 41 | 22
score on a scale | 70 [50 to 85] | 75 [55 to 80]

15. Secondary Outcome: Patient Health Questionnaire Scale (PHQ 8) Score at 90 Days
Description: The PHQ 8 has a range of 0 to 24 with 0 indicating no depression and 24 indicating severe depression.
Time Frame: 90 days post infusion
Population: Modified Intention To Treat population with PHQ 8 score available at 90 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 39 | 21
score on a scale | 4 [2 to 8] | 5 [2 to 10]

16. Secondary Outcome: Telephone Interview for Cognitive Status (TICS) Total Score at 30 Days Post Infusion
Description: The TICS has a range of 0 to 41 with a higher score indicating better cognitive status.
Time Frame: 30 days post infusion
Population: Modified Intent To Treat population with a TICS score at 30 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 34 | 18
score on a scale | 27 [19 to 32] | 21 [10 to 28]

17. Secondary Outcome: Telephone Interview for Cognitive Status (TICS) Total Score at 1 Year Post Infusion
Description: The TICS has a range of 0 to 41 with a higher score indicating better cognitive status.
Time Frame: 1 year post infusion
Population: Modified Intent To Treat population with a TICS score at 1 year
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 31 | 14
score on a scale | 31 [25 to 35] | 30 [23 to 33]

18. Secondary Outcome: Trail Making Test Score at 90 Days Post Infusion (Trail A)
Description: Both parts of the Trail Making Test consist of 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1 - 25, and the patient should draw lines to connect the numbers in ascending order. Reported in seconds needed to complete Trail A.
Time Frame: 90 days post infusion
Population: Modified Intent To Treat population with Trail A speed available
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 34 | 15
seconds | 78 [56 to 178] | 62 [44 to 90]

19. Secondary Outcome: Trail Making Test Score at 90 Days Post Infusion (Trail B)
Description: Both parts of the Trail Making Test consist of 25 circles distributed over a sheet of paper. In Part B, the circles include both numbers (1 - 13) and letters (A - L); as in Part A, the patient draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters. Reported in seconds needed to complete Trail B.
Time Frame: 90 days post infusion
Population: Modified Intent To Treat population with Trail B speed available
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 33 | 15
seconds | 278 [226 to 300] | 300 [142 to 300]

20. Secondary Outcome: Montreal Cognitive Assessment (MoCA) Score at 90 Days Post Infusion
Description: The MoCA has a range of 0 to 30 with lower scores indicating more severe cognitive impairment.
Time Frame: 90 days post infusion
Population: Modified Intent To Treat population with MoCA score available at 90 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 32 | 16
score on a scale | 21 [14.5 to 24.5] | 20 [8.5 to 24]

21. Secondary Outcome: Hopkins Verbal Learning Test-Revised (HVLT-R) Score at 90 Days Post Infusion
Description: The HVLT-R is a sum of three trials involving word recall. It has a total range of 0 to 36 with higher scores indicating better recall and greater cognition.
Time Frame: 90 days post infusion
Population: Modified Intent To Treat population with HVLT-R scores available at 90 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 33 | 16
score on a scale | 15 [9 to 21] | 12 [8.5 to 16]

22. Secondary Outcome: Short Form 36 Health Survey (SF-36) Scores at 90 Days Post Infusion
Description: For all sub-components (Physical Functioning, Role Limitations Due to Physical Health, Role Limitations Due to Emotional Problems, Energy/Fatigue, Emotional Well-being, Social Functioning, Pain, and General Health), a higher score indicates better health. Scales are standardized to obtain a score ranging from 0 to 100 and a mean score of 50 has been articulated as a normative value for all scales.
Time Frame: 90 days post infusion
Population: Modified Intent To Treat population with SF-36 scores available at 90 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 37 | 18
score on a scale
  Physical Functioning: number analyzed (Participants) | 37 | 17
  Physical Functioning | 30 [5 to 70] | 60 [5 to 75]
  Role Limitations Due to Physical Health: number analyzed (Participants) | 37 | 17
  Role Limitations Due to Physical Health | 0 [0 to 25] | 0 [0 to 25]
  Role Limitations Due to Emotional Problems: number analyzed (Participants) | 36 | 17
  Role Limitations Due to Emotional Problems | 66.7 [0 to 100] | 100 [0 to 100]
  Energy/Fatigue: number analyzed (Participants) | 37 | 17
  Energy/Fatigue | 55 [45 to 70] | 65 [45 to 85]
  Emotional Well-being: number analyzed (Participants) | 37 | 17
  Emotional Well-being | 72 [56 to 88] | 76 [64 to 84]
  Social Functioning: number analyzed (Participants) | 37 | 17
  Social Functioning | 62.5 [37.5 to 87.5] | 62.5 [50.0 to 87.5]
  Pain: number analyzed (Participants) | 37 | 17
  Pain | 67.5 [55 to 100] | 65 [42.5 to 80]
  General Health | 60 [50 to 75] | 70 [50 to 85]

23. Secondary Outcome: Controlled Oral Word Association Test (COWAT) Score at 90 Days Post Infusion
Description: The COWAT is a verbal fluency test in which participants are asked to say as many words as possible from a given category and in a specified timeframe (typically 60 seconds). Reported as the total number of words produced for F, A, and S. More words indicates better cognition.
Time Frame: 90 days post infusion
Population: Modified Intent To Treat population with COWAT score available at 90 days
Measure: Median (Inter-Quartile Range); unit: words
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 33 | 16
words | 14 [8 to 32] | 9.5 [6 to 22]

24. Secondary Outcome: Oral Symbol Digit Modalities Test (SDMT) Score at 90 Days Post Infusion
Description: The SDMT is a measure of processing speed wherein the participant is given 120 seconds to orally match symbols with digits as quickly as possible. Reported as the number of correct associations where a larger number indicates better cognition.
Time Frame: 90 days post infusion
Population: Modified Intent To Treat population with SDMT score available at 90 days
Measure: Median (Inter-Quartile Range); unit: associations
Arm/Group | Umbilical Cord Blood | Placebo
Number analyzed (Participants) | 30 | 15
associations | 13 [3 to 23] | 21 [8 to 34]

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Umbilical Cord Blood | Placebo
All-Cause Mortality (participants affected / at risk) | 4/52 | 1/27
Serious Adverse Events (participants affected / at risk) | 14/52 | 11/27
Other Adverse Events (participants affected / at risk) | 36/52 | 17/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Umbilical Cord Blood (N=52) | Placebo (N=27)
HEART FAILURE (Cardiac disorders) | 1 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 | 0
BRONCHIAL INFECTION (Infections and infestations) | 0 | 1
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
BULLOUS DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 1 | 0
COGNITIVE DISTURBANCE (Nervous system disorders) | 1 | 1
COLITIS (Gastrointestinal disorders) | 0 | 1
CONFUSION (Psychiatric disorders) | 1 | 0
DEATH NOS (General disorders) | 2 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 1
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ENDOCARDITIS INFECTIVE (Infections and infestations) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 2 | 2
FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 2 | 0
HYPOTENSION (Vascular disorders) | 1 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
INTRACRANIAL HEMORRHAGE (Nervous system disorders) | 1 | 0
ISCHEMIA CEREBROVASCULAR (Nervous system disorders) | 2 | 1
LEFT VENTRICULAR SYSTOLIC DYSFUNCTION (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 1
SEIZURE (Nervous system disorders) | 2 | 2
SEPSIS (Infections and infestations) | 0 | 1
SKIN INFECTION (Infections and infestations) | 1 | 0
STROKE (Nervous system disorders) | 1 | 2
THROMBOEMBOLIC EVENT (Vascular disorders) | 2 | 0
MUSCLE WEAKNESS RIGHT-SIDED (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Umbilical Cord Blood (N=52) | Placebo (N=27)
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
ANEMIA (Blood and lymphatic system disorders) | 3 | 4
ANOREXIA (Metabolism and nutrition disorders) | 2 | 3
ANXIETY (Psychiatric disorders) | 1 | 0
APNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
BACTEREMIA (Infections and infestations) | 1 | 0
CARDIAC DISORDERS - OTHER, SPECIFY (Cardiac disorders) | 0 | 1
CARDIAC TROPONIN T INCREASED (Investigations) | 0 | 2
CHEST PAIN - CARDIAC (Cardiac disorders) | 1 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
COGNITIVE DISTURBANCE (Nervous system disorders) | 5 | 1
CONCENTRATION IMPAIRMENT (Nervous system disorders) | 1 | 0
CONGENITAL, FAMILIAL AND GENETIC DISORDERS - OTHER (Congenital, familial and genetic disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 4
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 3
DELAYED ORGASM (Psychiatric disorders) | 0 | 1
DEPRESSION (Psychiatric disorders) | 5 | 5
DEVICE RELATED INFECTION (Infections and infestations) | 1 | 0
DIARRHEA (Gastrointestinal disorders) | 4 | 2
DIZZINESS (Nervous system disorders) | 0 | 1
DYSPEPSIA (Gastrointestinal disorders) | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 1 | 0
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 | 1
DYSURIA (Renal and urinary disorders) | 2 | 0
EDEMA LIMBS (General disorders) | 6 | 1
ENDOCRINE DISORDERS - OTHER, SPECIFY (Endocrine disorders) | 0 | 1
ESOPHAGITIS (Gastrointestinal disorders) | 1 | 0
EYE PAIN (Eye disorders) | 0 | 1
FALL (Injury, poisoning and procedural complications) | 6 | 3
FATIGUE (General disorders) | 2 | 0
FEVER (General disorders) | 2 | 1
FLATULENCE (Gastrointestinal disorders) | 1 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 5 | 4
HEART FAILURE (Cardiac disorders) | 0 | 1
HEMATURIA (Renal and urinary disorders) | 0 | 3
HEPATITIS B REACTIVATION (Infections and infestations) | 1 | 0
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 3 | 0
HYPERKALEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERNATREMIA (Metabolism and nutrition disorders) | 2 | 1
HYPERTENSION (Vascular disorders) | 6 | 0
HYPERURICEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPOKALEMIA (Metabolism and nutrition disorders) | 3 | 5
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPONATREMIA (Metabolism and nutrition disorders) | 2 | 1
HYPOTENSION (Vascular disorders) | 5 | 2
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ILEUS (Gastrointestinal disorders) | 1 | 0
INSOMNIA (Psychiatric disorders) | 4 | 3
INTRACRANIAL HEMORRHAGE (Nervous system disorders) | 0 | 1
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 1 | 0
ISCHEMIA CEREBROVASCULAR (Nervous system disorders) | 2 | 0
LEFT VENTRICULAR SYSTOLIC DYSFUNCTION (Cardiac disorders) | 1 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 7 | 1
LUNG INFECTION (Infections and infestations) | 4 | 1
MENORRHAGIA (Reproductive system and breast disorders) | 0 | 1
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIF (Metabolism and nutrition disorders) | 4 | 3
MUCOSITIS ORAL (Gastrointestinal disorders) | 1 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 4 | 0
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 12 | 4
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1 | 1
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 | 0
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 3 | 2
PERSONALITY CHANGE (Psychiatric disorders) | 1 | 0
PLATELET COUNT DECREASED (Investigations) | 1 | 0
PROSTATIC OBSTRUCTION (Reproductive system and breast disorders) | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 2 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 2 | 1
REPRODUCTIVE SYSTEM AND BREAST DISORDERS - OTHER, (Reproductive system and breast disorders) | 1 | 0
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - (Respiratory, thoracic and mediastinal disorders) | 0 | 1
SEIZURE (Nervous system disorders) | 3 | 2
SINUS BRADYCARDIA (Cardiac disorders) | 1 | 0
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 1
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SP (Skin and subcutaneous tissue disorders) | 1 | 0
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 2 | 1
SPASTICITY (Nervous system disorders) | 5 | 0
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 | 4
URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 2
URINARY TRACT INFECTION (Infections and infestations) | 5 | 5
URINE OUTPUT DECREASED (Investigations) | 0 | 1
VAGINAL INFECTION (Infections and infestations) | 2 | 2
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 3 | 0
INJURY, POISONING AND PROCEDURAL COMPLICATIONS - OTHER (Injury, poisoning and procedural complications) | 1 | 0
PAIN (General disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT03004976/Prot_SAP_000.pdf